CLINICAL TRIAL: NCT05568667
Title: Pilot Study to Improve Primary Prevention of Colorectal Cancer by Motivational and Community-based Approaches, According to Individual Risk Level, in People Undergoing Colonoscopy
Brief Title: Improve Colorectal Cancer Prevention by Motivational and Community-based Approaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRECÔTION
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2023-03

CONDITIONS: Colorectal Cancer Prevention
MeSH Terms: interventions — AIEOP acute lymphoblastic leukemia protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Risk sub-group (Experimental): 1. st sub-grouup : Low risk to develop a CRC
  2. nd sub-group : Moderate risk to develop a CRC
  3. rd sub-group : High risk to develop a CRC
  Interventions: Behavioral: Low risk; Behavioral: Moderate risk; Behavioral: High risk

INTERVENTIONS:
Behavioral: Low risk — * remote support in physical activity and nutrition via digital media
  * monthly collective physical activity sessions
  * logbook
Behavioral: Moderate risk — * remote support in physical activity and nutrition via digital media
  * monthly collective physical activity sessions
  * one collective health education session
  * logbook
Behavioral: High risk — * remote support in physical activity and nutrition via digital media
  * monthly collective physical activity sessions
  * one collective health education session
  * 3 individual sessions of motivational coaching
  * connected watch
  * logbook

SUMMARY:
It has been estimated that 19,000 Colorectal Cancers (CRC) could be prevented each year in France by changing individual risk behaviours (sedentary lifestyle, overweight, diet, alcohol). The cancer screening appears to be an opportune moment for health promotion and to inform about CRC risk factors.

The PRECÔTION study proposes an innovative scheme based on informative, motivational and community-based approaches. The objectives are to take advantage of patients' visits for colonoscopy to raise awareness and initiate individual prevention actions according to their own risk in order to modify individual risk behaviour.

Patients who come for a colonoscopy at the Centre Léon Bérard and who are negative (80% of cases) will benefit from an evaluation to identify their individual risk factors, determine their level of risk level for CRC and their motivation to change their behaviour.

Participants with a low level of risk will receive remote support in physical activity and nutrition via digital media based on a motivational approach. Participants will be proposed a monthly collective physical activity session, which will allow them to interact with each other and develop a community approach. Participants with an intermediate level of risk will be offered a collective health education session, in addition to the the support offered to participants with a low level of risk. Participants with a high level of risk will receive, in addition to the the support offered to participants with an intermediate level of risk, an individual motivational coaching and a connected watch. A logbook will also be given to all participants to accompany them on the different tools, especially for monitoring their goals.

The PRECÔTION study aims to evaluate these tools as innovative means of prevention before evaluate their effectiveness on a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* I1. Adult aged ≤ 80 years,
* I2. Having undergone in the month prior to inclusion a colonoscopy for CRC screening, with a negative result,
* I3. Willing to be involved throughout the study,
* I4. Able to practice a adapted physical activity (APA) certified by a medical certificate issued by the referring oncologist or the clinical investigator,
* I5. Using a own smartphone, a tablet or a PC with Internet connexion,
* I6. Having a valid health insurance affiliation,
* I7. Having dated and signed an informed consent form,
* I8. Able to read, write and understand French.

Exclusion Criteria:

* NI1. Presence of a primary cancer (other than in situ cancer of any location and/or basal cell skin cancer) - NB : people in complete remission from a previous cancer may be included,
* NI2. With a contraindication to pratice physical activity (e.g. uncontrolled hypertension, uncontrolled heart disease),
* NI3. Severe undernutrition (HAS) (i.e. weight loss ≥ 10% in 1 month or ≥ 15% in 6 months or ≥ 15% compared to usual weight or body mass index ≤ 17 kg/m² for a person < 70 ans or body mass index < 20 kg/m² for a person ≥ 70 ans)
* NI4. Unable to be followed for medical, social, family, geographical or psychological reasons throughout the study,
* NI5. Deprived of liberty by judicial or administrative decision,
* NI6. Concurrent participation in another PA or nutrition study,
* NI7. (For women) Pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Assessment of the programme feasability | Month 6
  Participation rate at each modality of the programme

SECONDARY OUTCOMES:
Assessment of the programme acceptability | Month 6
  Participation rate to the study (number of participants/number of eligible persons)
Assessment of the programme acceptability | Month 6
  Satisfaction, assessed by a Likert scale on a self-administered questionnaire
Assessment of the programme observance | Month 6
  Evaluate the observance to the whole programme, for each subgroup
Assessment of the evolution of lifestyle | Month 6
  World Cancer Research Fund international questionnaire Score : from 0 (worse score) to 7 (better score)
Assessment of the physical activity level change | Month 6
  Evaluate the effects on physical activity level using the IPAQ
Assessment of the evolution on CRC risk factors knowledge | Month 6
  Self-administered questionnaire (questionnaire specially designed for the study, no titlle) Score : from 0 (worse score) to 9 (better score)

CONTACTS AND LOCATIONS:
Overall Officials: Anne CATTEY-JAVOUHEY, MD, PhD, Principal Investigator — Centre Leon Berard
Locations (1):
- Centre Léon Bérard (CLB), Lyon, France

IPD SHARING:
Plan to Share IPD: No